CLINICAL TRIAL: NCT06155123
Title: High-density EEG Evaluation of Functional Connectivity Changes in Migraine Patients Receiving Advanced Preventive Therapies (Anti-CGRP mAbs)
Brief Title: HD-EEG Connectivity Changes in Migraine Patients Undergoing Treatment With Anti-CGRP mAbs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HD-EEG in mAbs
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Migraine Disorders; Chronic Migraine; Episodic Migraine
Keywords: migraine; anti CGRP mAbs; HD EEG; brain connectivity; resting state networks
MeSH Terms: conditions — Migraine Disorders | interventions — Ligands

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFEM or CM treated with mAbs: Patients with high frequency episodic or chronic migraine undergoing treatment with monoclonal antibodies directed against calcitonin gene related peptide pathway
  Interventions: Drug: Monoclonal antibody targeting the CGRP pathway (ligand or receptor) (mAbs)
- Healthy Controls: Group of healthy controls comparable for demographic features

INTERVENTIONS:
Drug: Monoclonal antibody targeting the CGRP pathway (ligand or receptor) (mAbs) — Monthly or quarterly mAbs administration for a year
  Groups: HFEM or CM treated with mAbs

SUMMARY:
Migraine is a leading cause of disability with an estimated prevalence of 12% in Europe. The headache field witnessed a breakthrough since the introduction of specific preventive therapies which proved effective and well tolerated, namely the monoclonal antibodies directed against the Calcitonin Gene Related Peptide (CGRP) pathway (mAbs). Their mechanism of action is still debated. Several Authors claimed that, despite the site of action is peripheral (namely outside of the blood brain barrier), the resulting action may take place at central level. Another valuable hypothesis is that the clinical modifications resulting from mAbs treatment may induce functional modulation of several brain areas.

With these premises, the primary aim of the study is to evaluate changes in functional connectivity in patients undergoing preventive mAbs treatment using high density EEG.

DETAILED DESCRIPTION:
Electroencephalogram (EEG) is widely available as a powerful mean to non-invasively study brain connectivity features in migraine patients. High density EEG, by means of a minimum of 64 up to 256 electrodes, enables to record electrical brain activity with high spatial resolution. Through the analysis of brain oscillations across different frequency bands (from alpha to delta), it can evaluate sensory, pain processing and information integration, contributing to a better definition of baseline features and to detect potential markers or predictors for therapeutic interventions in an era addressed to precision medicine.

Previous neurophysiological studies focused on EEG and to assess functional connectivity or spectral analysis in migraine patients. Conventional studies found higher slow wave activity (predominantly theta) in the interictal phase and higher excitability in the visual cortex during visual aura.

In 2016 a resting state study showed a predominance of low frequency bands in the ictal phase. The interictal and ictal phases patients also presented a diffuse lower coherence, suggesting low functional connectivity. Furthermore, an altered spatial connectivity for lower alpha-band activities was found in the interictal phases during sensory stimulation by means of HD-EEG, suggesting a thalamocortical dysrhythmia.

Nowadays, targeted preventive migraine therapies are available, namely monoclonal antibodies directed against the Calcitonin Gene Related Peptide (CGRP) pathway (mAbs). They demonstrated high efficacy and tolerability in both chronic and episodic migraine. Despite their peripheral site of action (outside of the blood brain barrier), the resulting action may take place at central level or determine clinical modifications leading to a functional modulation of several brain areas.

The primary aim of the study is to evaluate changes in functional connectivity in patients undergoing preventive mAbs treatment using HD- EEG and eventual connectivity differences between Responders and Non-Responders.

Study design:

Patients will undergo visits planned at baseline (T0) and quarterly (T3-T6) during which clinical data is collected and an HD-EEG is performed. Healthy controls will undergo EEG registration once.

HD-EEG registration:

The investigators will randomly acquire 4 recordings (6 minutes each) in resting-state condition, 2 with opened eyes, and 2 with closed eyes.

Resting state FC will be analyzed among six resting state networks (Default mode network, Dorsal attention network, Ventral attention network, Language network , Somatomotor network and Visual network) in the following frequency bands: alfa 8-12 Hz, beta 13-30 Hz, gamma 31-80 Hz, theta 4-7 Hz. delta 1-3 Hz.

Acquisition parameters will be: High-Pass: 0.5 Hz; Low-Pass: 100 Hz; Notch: 50 Hz. For analysis of HD-EEG data, the investigators will use a tailored analysis pipe-line that was previously developed and validated to reconstruct neural sources from cortical/subcortical gray matter. EEG signals will be band-pass filtered (1-80 Hz) and down-sampled at 250 Hz. Biological artifacts will be rejected using Independent Component Analysis (ICA). EEG signals will be referenced with a customized version of the Reference Electrode Standardization Technique (REST). A matrix will estimate the relationship between the measured scalp potentials and the dipoles corresponding to brain sources. Sources reconstruction will be performed with the exact low-resolution brain electromagnetic tomography (eLORETA) algorithm

Statistical plan:

The sample size was computed with the freeware online platform www.openepi.com. As few studies focused on functional connectivity evaluation in migraine, with no studies analyzing longitudinal changes during a specific treatment, the sample size analysis was based on the work of Bjork. The investigators thus considered as clinically meaningful a difference between groups in the theta relative power band equal to 0.04 (±0.04). Considering a two-tailed t-test for the comparison with confidence interval 95%; power: 80%, the minimum suggested sample size was 20 subjects for CM group and 20 subjects for HFEM group.

A preliminary normality analysis will be performed to decide whether to use parametric or non-parametric methods, through Shapiro Wilk test.

Numerical variables will be described as mean and standard deviation (or median and quartiles if appropriate), categorical variables as raw numbers and percentages.

Functional connectivity analyses will be conducted for separate bands and eyes closed registration.

ELIGIBILITY:
Inclusion Criteria:

* Episodic or chronic migraine diagnosis according to ICHD-3 criteria
* Indication to BoNT-A or mAbs treatment according to AIFA criteria
* Brain MRI performed within 24 months from enrolment

Exclusion Criteria:

* Previous or actual history of epilepsy
* Diagnosis of dementia o mental retardation
* Diagnosis of psychiatric illness according to Diagnostic and Statistical Manual of Mental Disorders V
* Other concomitant type of headache (except for sporadic tension type headache)
* Chronic pain conditions
* Pregnancy or breastfeeding
* Concomitant use of electrical stimulators, pace-makers, metallic clips or other metallic foreign bodies
* Previous head surgery
* Ongoing neuroactive prevention therapies or other drugs, or psicoactive substances possibly interfering with EEG recording (eg benzodiazepines)
* Other conditions possibly influencing EEG recording
* Brain anomalies detected on MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic and high frequency episodic migraine attending the outpatient clinic of the Headache Science & Neurorehabilitation Center of the IRCCS Mondino Foundation (Pavia, Italy).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Differences in absolute functional connectivity values (continuous variable, without unit of measurement) in resting state networks (RSN-FC) in migraine group across 6 months of mAbs treatment. | Baseline (T0) - 3 months of mAbs treatment (T3) - 6 months of mAbs treatment (T6)
  To compare HD-EEG functional connectivity in migraine patients across 6 months of mAbs treatment
Differences in absolute functional connectivity values (continuous variable, without unit of measurement) in Responders vs. Non-Responders across 6 months of mAbs treatment | Baseline (T0) - 3 months of mAbs treatment (T3) - 6 months of mAbs treatment (T6)
  To compare HD-EEG functional connectivity in Responders (those who achieved a reduction of Monthly migraine days > / = 50% compared to T0) vs. Non-Responders across 6 months of mAbs treatment

SECONDARY OUTCOMES:
Baseline differences in absolute functional connectivity values (continuous variable, without unit of measurement) among patients with a baseline diagnosis of HFEM vs. CM vs. healthy controls | Baseline (T0)
  To compare HD-EEG functional connectivity among HFEM group (patients with > / = 8 MMDs at T0) vs. CM group (patients with > / = 15 MMDs at T0) vs. healthy controls
Baseline differences in absolute functional connectivity values (continuous variable, without unit of measurement) in Responders vs. Non-Responders | Baseline (T0)
  To compare HD-EEG functional connectivity in Responders (those who achieved a reduction of Monthly migraine days > / = 50% vs. T0) vs. Non-Responders at baseline

OTHER OUTCOMES:
Differences in monthly migraine days across 6 months of mAbs treatment (continuous variable) | Baseline (T0) - six months of mAbs treatment (T6)
  To evaluate differences in monthly migraine days across 6 months of mAbs treatment
Differences in monthly headache days across 6 months of mAbs treatment (continuous variable) | Baseline (T0) - six months of mAbs treatment (T6)
  To evaluate differences in monthly headache days across 6 months of mAbs treatment
Differences in monthly days of acute drugs consumption across 6 months of mAbs treatment (continuous variable) | Baseline (T0) - six months of mAbs treatment (T6)
  To evaluate differences in monthly days of acute drugs consumption across 6 months of mAbs treatment
Differences in monthly doses of acute drugs consumption across 6 months of mAbs treatment (continuous variable) | Baseline (T0) - six months of mAbs treatment (T6)
  To evaluate differences in monthly doses of acute drugs consumption across 6 months of mAbs treatment
Differences in disability in migraine group across 6 months of mAbs treatment (continuous variable ranging from 0-270) | Baseline (T0) - six months of mAbs treatment (T6)
  To evaluate differences in Migraine Disability Assessment Score (MIDAS) Questionnaire across 6 months of mAbs treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Science & Neurorehabilitation Center, Pavia, Italy

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Bjork MH, Stovner LJ, Engstrom M, Stjern M, Hagen K, Sand T. Interictal quantitative EEG in migraine: a blinded controlled study. J Headache Pain. 2009 Oct;10(5):331-9. doi: 10.1007/s10194-009-0140-4. Epub 2009 Aug 25. PMID 19705061
- [Background] Coppola G, Di Lorenzo C, Parisi V, Lisicki M, Serrao M, Pierelli F. Clinical neurophysiology of migraine with aura. J Headache Pain. 2019 Apr 29;20(1):42. doi: 10.1186/s10194-019-0997-9. PMID 31035929
- [Background] de Tommaso M, Trotta G, Vecchio E, Ricci K, Siugzdaite R, Stramaglia S. Brain networking analysis in migraine with and without aura. J Headache Pain. 2017 Sep 29;18(1):98. doi: 10.1186/s10194-017-0803-5. PMID 28963615
- [Background] Cao Z, Lin CT, Chuang CH, Lai KL, Yang AC, Fuh JL, Wang SJ. Resting-state EEG power and coherence vary between migraine phases. J Headache Pain. 2016 Dec;17(1):102. doi: 10.1186/s10194-016-0697-7. Epub 2016 Nov 2. PMID 27807767
- [Background] Chamanzar A, Haigh SM, Grover P, Behrmann M. Abnormalities in cortical pattern of coherence in migraine detected using ultra high-density EEG. Brain Commun. 2021 Apr 2;3(2):fcab061. doi: 10.1093/braincomms/fcab061. eCollection 2021. PMID 34258580
- [Background] Semprini M, Bonassi G, Barban F, Pelosin E, Iandolo R, Chiappalone M, Mantini D, Avanzino L. Modulation of neural oscillations during working memory update, maintenance, and readout: An hdEEG study. Hum Brain Mapp. 2021 Mar;42(4):1153-1166. doi: 10.1002/hbm.25283. Epub 2020 Nov 17. PMID 33200500
- [Background] Aoki Y, Ishii R, Pascual-Marqui RD, Canuet L, Ikeda S, Hata M, Imajo K, Matsuzaki H, Musha T, Asada T, Iwase M, Takeda M. Detection of EEG-resting state independent networks by eLORETA-ICA method. Front Hum Neurosci. 2015 Feb 10;9:31. doi: 10.3389/fnhum.2015.00031. eCollection 2015. PMID 25713521